CLINICAL TRIAL: NCT03705312
Title: EValuation of Outcomes of Transcatheter Mitral Valve Repair for the Treatment of Low Ejection Fraction and Moderate Functional Mitral ValvE Regurgitation In Heart Failure
Brief Title: MitraClip for the Treatment of Moderate Functional Mitral Regurgitation: EVOLVE-MR
Acronym: EVOLVE-MR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montreal Heart Institute (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-2458
Record Dates: First submitted 2018-08-04; First posted 2018-10-15 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2018-10

CONDITIONS: Mitral Regurgitation; Heart Failure; Mitral Valve Regurgitation Due to Cardiomyopathy (Disorder)
Keywords: mitral regurgitation; transcatheter mitral valve repair
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to medical treatment or intervention with the MitraClip device
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Guideline-directed medical therapy (Placebo Comparator): Standard guideline-directed medical treatment for heart failure
  Interventions: Other: Guideline-directed medical therapy
- Transcatheter Mitral valve repair (Experimental): MitraClip treatment
  Interventions: Device: Transcatheter mitral valve repair

INTERVENTIONS:
Device: Transcatheter mitral valve repair — Transcatheter mitral valve repair performed using the MitraClip device
  Other Names: MitraClip
  Arms: Transcatheter Mitral valve repair
Other: Guideline-directed medical therapy — Standard medical therapy for heart failure as recommended by HF guidelines
  Arms: Guideline-directed medical therapy

SUMMARY:
This study evaluates the addition of transcatheter mitral valve repair with the MitraClip device to medical treatment in patients with heart failure and moderate functional mitral regurgitation to determine the impact of left ventricular remodelling and patients' functional capacity.

DETAILED DESCRIPTION:
Moderate mitral regurgitation in patients with LV dysfunction is associated with increased risk of death and hospitalizations for heart failure (HF) and leads to progressive remodelling of an already damaged left ventricle. Medical therapies and cardiac resynchronization therapy (CRT) have demonstrated favourable effects on LV remodelling in heart failure patients.

Given the benefits and safety of transcatheter mitral valve repair with the MitraClip device in severe MR, it is conceivable that this technology could also be safely used in those with moderate MR to reduce mitral regurgitation, improve symptoms and result in LV remodelling. At present, the optimal treatment strategy for heart failure patients and moderate (2+, 2-3+) mitral regurgitation is uncertain therefore the EVOLVE-MR study proposes to evaluate transcatheter mitral valve repair with the MitraClip in such patients to study the effects on LV remodelling and functional capacity.

EVOLVE-MR is a randomized study of MitraClip and medical therapy in symptomatic heart failure patients with moderate (2+, 2-3+) secondary mitral regurgitation. The objective of this study is to determine the impact of both therapies on left ventricular remodelling and functional capacity of the target patient population.

ELIGIBILITY:
Inclusion Criteria:

* Moderate functional mitral regurgitation (2+, 2-3+)
* Left ventricular ejection fraction >20%
* LVEDV 75-110 ml/m2
* Symptomatic heart failure (NYHA Class II-IV)

Exclusion Criteria:

* Left ventricular ejection fraction < 20%
* Severe functional mitral regurgitation
* Recent coronary artery bypass graft surgery (CABG)
* Untreated significant coronary artery disease
* Mitral valve area < 4.0cm2
* Severe pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular diastolic remodelling | 12 months
  Change in indexed left ventricular diastolic volume (LVEDV)
Functional capacity as measured by 6 minute walk test | 12 months
  Change in distance walked on six-minute walk test

SECONDARY OUTCOMES:
Mitral regurgitation Severity (RV) | 12 months
  Change in mitral regurgitant volume
Mitral regurgitation Severity (EROA) | 12 months
  Change in effective regurgitant orifice area
Quality of Life Measurement | 12 months
  Change in indices of quality of life as measured by Kansas City Cardiomyopathy Questionnaire. The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Anita W Asgar, MD, Principal Investigator — Montreal Heart Institute; Anique Ducharme, MD, Principal Investigator — Montreal Heart Institute; Jean L Rouleau, MD, Study Chair — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided